CLINICAL TRIAL: NCT00075140
Title: Family Health After Predictive Huntington Disease Testing
Brief Title: Family Health After Predictive Huntington Disease (HD) Testing
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Janet K. Williams, PhD, RN, FAAN, University of Iowa
Other Study IDs: 1R01NR007970-01 (NIH)
Record Dates: First submitted 2004-01-02; First posted 2004-01-05 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Huntington Disease
Keywords: Patient Care Management; Family; Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All Participants hav a family member with Huntington Disease
  Interventions: Genetic: Mutation in the gene

INTERVENTIONS:
Genetic: Mutation in the gene

SUMMARY:
The purpose of this study is to identify health management concerns and needs of family members of asymptomatic and symptomatic persons with mutation in the gene for Huntington Disease (HD).

DETAILED DESCRIPTION:
This is an observational study with three phases. In Phase 1, focus groups consisting of family members of persons with HD Gene mutation will be conducted and data collected to be analyzed through content analysis to identify salient themes and key issues. In Phase 2, a survey instrument will be developed and field-tested in order to describe the health care needs, management strategies, and needs for health and social services of relative/significant others of asymptomatic and symptomatic persons with the mutation in the gene for HD.

In Phase 3, the survey will be distributed to family members of asymptomatic and symptomatic persons with mutation in the gene for HD and frequencies and comparisons of survey responses according to respondent characteristics will be reported.

ELIGIBILITY:
* Family members of asymptomatic and symptomatic persons with mutation in the gene for Huntington Disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Family members or significant others, age 14 or older, of persons who 1) have received a positive result from predictive testing for a mutation in the HD gene, 2) are symptomatic and living at home, and 3) are symptomatic and are living in a long-term care institution were the population of interest for this study.
Sampling Method: Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2001-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Impact of a positive HD test or presence of HD on a family members perceptions of: health problems, emotional and functional health status, resources/strategies for managing problems, helpfulness, and services needed to help family members cope. | Over 6 yr span

SECONDARY OUTCOMES:
Describe the health care needs, management strategies, and needs for health and social services of a broader sample of relatives/significant others in families in which a person has a gene mutation for HD. | Over 6 yr span

CONTACTS AND LOCATIONS:
Overall Officials: Janet K Williams, PhD, RN, FAAN, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa College of Nursing, Iowa City, Iowa, United States